CLINICAL TRIAL: NCT07117955
Title: Treatment of Peyronie's Disease With Platelet-Rich Plasma: A Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Platelet-Rich Plasma for Peyronie's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Mikael Heering, Medical Doctor, PhD-student, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-24019622
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Peyronies Disease
Keywords: Andrology; Platelet-Rich Plasma; Penile induration; PRP
MeSH Terms: conditions — Penile Induration | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The participant and the investigator/treating doctor will be masked. The syringes will be covered. Only the care provider who prepare the PRP will not be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platelet Rich Plasma (PRP) (Experimental)
  Interventions: Other: Autologous Platelet Rich Plasma
- Saline Solution (Placebo) (Placebo Comparator)
  Interventions: Other: Saline solution

INTERVENTIONS:
Other: Autologous Platelet Rich Plasma — 6 mL PRP intralesional injections will be administered. After the injections, participants will be instructed to perform penile stretching exercises daily until the next injection and to continue these exercises after the final injection until the 3-month follow-up.
  Other Names: PRP
  Arms: Platelet Rich Plasma (PRP)
Other: Saline solution — 6 mL saline solution intralesional injections will be administered. After the injections, participants will be instructed to perform penile stretching exercises daily until the next injection and to continue these exercises after the final injection until the 3-month follow-up.
  Other Names: Placebo
  Arms: Saline Solution (Placebo)

SUMMARY:
The purpose of this clinical trial is to evaluate the effects of Platelet-Rich Plasma (PRP) intralesional injections in men affected by Peyronie's disease (PD) in the fibrotic phase.

DETAILED DESCRIPTION:
The study protocol is structured such that participants, after being informed about the project and providing consent, will attend a baseline visit where relevant data will be collected from the participant, questionnaires, the patient's medical record, and through an objective examination. A total of 84 patients with Peyronie's disease will be included. Participants will be stratified based on the degree of penile curvature at baseline (30-60 degrees or >60 degrees) and randomized in a 1:1 ratio to receive either active treatment with Platelet-Rich Plasma (PRP) or placebo (saline). Subsequently, participants will attend weekly injection sessions for 3 weeks consisting of either PRP or saline in a randomized, double-blind manner. A follow-up visit will take place three months after the final injection for outcome assessment. Two additional long-term follow-up visits will be conducted at 6 and 12 months post-treatment. Analysis will then be conducted.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Be able to provide written informed consent
* Diagnosis of PD without active pain and without progressive curvature over the past 3 months (fibrotic phase).
* Penile curvature of 30-95 degrees
* Clearly palpable penile plaque

Exclusion Criteria:

* Erectile Dysfunction unresponsive to on-demand PDE5 inhibitors
* Hourglass malformation
* Severely calcified plaques where injection is considered unfeasible
* Intrapenile plaque
* History of priapism.
* History of penile fracture.
* Previous treatment for PD with injections and/or surgery.
* Antithrombotic therapy associated with a high risk of bleeding

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Degree Changes in Penile Curvature. | From enrollment to 12 months post intervention.
  Dominant curvature angles will be measured bedside in the outpatient clinic using a goniometer following intracavernosal administration of Alprostadil to ensure high quality and consistency. At the same visit, standardized photographs of the erect penis will be captured (in two plans) to support objective assessment. These procedures will be performed at baseline and at follow-up three months after the final injection.
  At the 6- and 12-months long-term follow-up visits, no pharmacological erection induction will be performed. Instead, penile curvature will be assessed based on standardized photographs of the participant's erection taken at home following detailed instructions, allowing evaluation of the durability of any treatment effect.

SECONDARY OUTCOMES:
Changes in Plaque Size | From enrollment to 12 months post intervention.
  Plaque size will be measured at baseline and 3, 6 and 12 months after the final injection using a ruler, calculated as the product of plaque length and width. Participants with more than two plaques or with significant plaque heterogeneity will not have plaque size measured and will be excluded from these analyses but may still participate in the study.
Changes in the Peyronie's Disease Questionnaire (PDQ) | From enrollment to 3 months post intervention.
  The Peyronie's Disease Questionnaire (PDQ) is a 15-question self-reported survey that measures the impact and severity of Peyronie's disease (PD) symptoms in 3 domains, including psychological and physical symptoms, penile pain and symptom bother.
  Higher domain scores indicate a greater negative impact. The range of scores for each domain is 0 to 24 for PD psychological and physical symptoms, 0 to 30 for penile pain and 0 to 16 for PD symptom bother.
  The participants will complete the survey at baseline and 3, 6 and 12 months after the final injection.
Changes in the Erection Hardness Score (EHS) | From enrollment to 12 months post intervention.
  The participants will rate the hardness of their erection via the single-item Likert scale EHS, at baseline and 3, 6 and 12 months after the final injection. The scale is from 0-4. 0 is no erection, the higher the score the better erection.
Changes in the Major Depression Inventory (MDI) | From enrollment to 12 months post intervention.
  The Major Depression Inventory (MDI) is a patient-reported outcome measure to assist with diagnosing and evaluation of the severity of a patient's depression.
  The MDI score ranges from 0 to 50, where 0 represents no depression symptoms and 50 represents the most severe depression symptoms.
  The participants will complete the MDI questionnaire at baseline and 3, 6 and 12 months after the final injection.
  The MDI is included due to previously described associations between Peyronie's disease and depression. The data may be used to assess the impact of disease progression on potential depressive symptoms.
The Ability to Engage in Sexual Intercourse (question) | From enrollment to 12 months post intervention.
  The participants will be assessed at baseline and 3, 6 and 12 months after the final injection regarding their ability to engage in sexual intercourse. This will be assessed by asking participants a single binary question: whether they are able to engage in sexual intercourse (yes or no).
Preference for Surgical Intervention (question) | From enrollment to 12 months post intervention.
  The participants will be inquired about their preference for surgical intervention in relation to the current penile curvature at baseline and 3, 6 and 12 months after the final injection. This will be assessed by asking participants a single binary question: whether they wish to undergo surgery given their current curvature (yes or no).
Changes in Global Assessment Scale Questionnaire | From 3 to 12 months post intervention.
  The participants will complete a Global Assessment Scale Questionnaire regarding overall treatment satisfaction at the 3-, 6- and 12 months follow-up after the final injection.
  The questionnaire consists of a single question regarding the participants' overall satisfaction with the treatment, to be answered on a scale from 1 to 5. A higher value indicates greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel M. Fode, Professor, MD, Ph.d., Principal Investigator — Herlev and Gentofte University Hospital
Locations (1):
- Herlev and Gentofte University Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No